CLINICAL TRIAL: NCT03143764
Title: Bicycle Usage and Cardiorespiratory Fitness Among Inactive Adults Provided With Electrically Assisted Bicycles
Brief Title: Cardiorespiratory Fitness Using Electrically Assisted Bicycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: The GC Rieber Funds (Unknown); Bergen Council (Other); Helse Stavanger HF (Other Government); Kristiansand Zoo and Amusement park (Unknown); National Oilwell Varco Norway AS (Unknown); General Practitioner-scholarship from the Norwegian Medical Association. (Unknown); Department of Global Public Health and Primary Care, University of Bergen (Unknown); Department of Education and Sports Science, University of Stavanger (Unknown); Department of Sports and Physical Activity, Bergen University College (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UBergenElsykkel
Record Dates: First submitted 2017-04-21; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Transportation

STUDY DESIGN:
Intervention Model Description: Inactive employees in a selection of public and private corporations in three Norwegian cities were invited to participate. Inclusion criteria were: a desire to cycle to work, residence more than 3km from the workplace, and not physically active according to guidelines. There were 25 participants in the study and we provided them all with electrically assisted bicycles fitted with GPS bike computers to record usage. The participants were followed for three to eight months, 226 days on average
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Commuting with electrically assisted bicycles — 25 participants were provided with electrically assisted bicycles fitted with GPS bike computers to record usage

SUMMARY:
This study aimed to examine cycling time and distance when inactive subjects were provided with electrically assisted bicycles, and secondly, to examine changes in cardiorespiratory fitness.

DETAILED DESCRIPTION:
Method: Inactive employees in a selection of public and private corporations in three Norwegian cities were invited to participate. Inclusion criteria were: a desire to cycle to work, residence more than 3km from the workplace, and not physically active according to guidelines. There were 25 participants in the study and we provided them all with electrically assisted bicycles fitted with GPS bike computers to record usage. The participants were followed for three to eight months, 226 days on average. Measures of maximal oxygen uptake were performed before and after the intervention. Demographic characteristics and prior transportation habits were reported in a questionnaire at baseline.

ELIGIBILITY:
Inclusion Criteria:

-a desire to cycle to work, residence more than 3km from the workplace, and not physically active according to guidelines

Exclusion Criteria:

-

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-06-15 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
examine cycling time | 12 months
  when inactive subjects were provided with electrically assisted Bicycles for 12 months
examine cycling distance | 12 months
  when inactive subjects were provided with electrically assisted Bicycles for 12 months

SECONDARY OUTCOMES:
examine changes in cardiorespiratory fitness | 12 months
  Measurements of V02 max pre- post

CONTACTS AND LOCATIONS:
Locations (3):
- Norway (3):
  - Department of Global Public Health and Primary Care, University of Bergen, Bergen
  - Department of Public Health, Sport and Nutrition, University of Agder, Kristiansand
  - Department of Education and Sports Science, University of Stavanger, Stavanger

IPD SHARING:
Plan to Share IPD: No